CLINICAL TRIAL: NCT00748098
Title: Study RXP110908, a Polysomnography Study of GSK1838262 (XP13512) Extended Release Tablets Versus Placebo in the Treatment of Restless Legs Syndrome (RLS) and Associated Sleep Disturbance
Brief Title: Polysomnography Study of GSK1838262 Extended Release Tablets Versus Placebo in RLS and Associated Sleep Disturbance
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: XenoPort, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RXP110908
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Results first posted 2011-05-18 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-01

CONDITIONS: Restless Legs Syndrome; Restless Legs Syndrome (RLS)
Keywords: PSG; Restless Legs Syndrome; gabapentin enacarbil; XP13512; GSK1838262; sleep disturbance; RLS; polysomnography
MeSH Terms: conditions — Restless Legs Syndrome; Parasomnias | interventions — 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK1838262:placebo (Other): GSK1838262 extended release tablets for Treatment Period 1 followed by Placebo for Treatment Period 2
  Interventions: Drug: Placebo
- Placebo:GSK1838262 (Other): Placebo for Treatment Period 1 followed by GSK1838262 for Treatment Period 2
  Interventions: Drug: GSK1838262 Extended Release Tablets

INTERVENTIONS:
Drug: GSK1838262 Extended Release Tablets — GSK1838262 extended release tablets
  Other Names: XP13512; gabapentin enacarbil
  Arms: Placebo:GSK1838262
Drug: Placebo — Placebo
  Arms: GSK1838262:placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of GSK1838262 extended release tablets in the treatment of patients with Restless Legs Syndrome and associated sleep disturbance.

DETAILED DESCRIPTION:
Double-blind, multi-center, placebo-controlled, 2-period crossover study which assessed the efficacy and safety of gabapentin enacarbil (GEn; GSK1838262; XP13512) extended release tablets in adults with Restless Legs Syndrome (RLS)-associated sleep disturbance. One hundred thirty-six (136) adult subjects with RLS-associated sleep disturbance and periodic limb movements (PLM) were randomized from 23 centers in the United States. Subjects who met all eligibility criteria were randomized to receive a treatment sequence of GEn:placebo or placebo:GEn. Investigational product was taken with food at approximately 5pm. Investigational product was dosed as 600mg/day x3 days followed by 1200mg/day x25 days for each 4-week treatment period. There was a 1-week taper at 600mg after each treatment period followed by a 1-week washout between treatments. Polysomnography (PSG) was used to objectively evaluate changes in sleep and PLMs.

ELIGIBILITY:
Inclusion criteria:

* Provided written informed consent.
* Diagnosed with primary RLS using the International RLS Study Group Diagnostic Criteria with a total score of 15 or greater on the International RLS (IRLS) Rating Scale and significant sleep disturbance indicated on Item 4 of the IRLS rating scale.
* Have history of RLS symptoms at least 15 nights/month.
* Minimum average of 15 Periodic Limb Movements during Sleep per hour (measured using actigraphy).

Exclusion criteria:

* Secondary RLS
* Primary sleep disorder
* Sleep apnea
* Have any medical conditions that may impact efficacy assessments or that may present a safety concern.
* Pregnant or lactating or women of child-bearing potential who are not practicing an acceptable method of birth control.
* Use of any prohibited medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2008-10; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (23):
- United States (23):
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Hallandale, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Crestview Hills, Kentucky
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Chevy Chase, Maryland
  - GSK Investigational Site, Brighton, Massachusetts
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, West Seneca, New York
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Dublin, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Walla Walla, Washington

REFERENCES:
- [Background] Calloway M, Bharmal M, Hill-Zabala C, Allen R. Development and validation of a subjective post sleep diary (SPSD) to assess sleep status in subjects with restless legs syndrome. Sleep Med. 2011 Aug;12(7):704-10. doi: 10.1016/j.sleep.2010.09.020. Epub 2011 Jul 5. PMID 21733752

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Followed by GEn 1200 mg/Day: Participants randomized to matching placebo administered once daily with food at 5 pm during the 28-day First Treatment Intervention Period and the 7-day First Taper Period. No treatment was given during the 7-day Washout. Gabapentin enacarbil (GEn) 1200 mg/day administered once daily with food at 5 pm during the 28-day Second Treatment Intervention Period (Days 1-3, 600 mg). GEn 600 mg administered once daily with food at 5 pm during the 7-day Second Taper Period. No treatment was given during Follow-up.
- GEn 1200 mg/Day Followed by Placebo: Participants randomized to GEn 1200 mg/day administered once daily with food at 5 pm during the 28-day First Treatment Intervention Period (Days 1-3, 600 mg). GEn 600 mg administered once daily with food at 5 pm during the 7-day First Taper Period. No treatment was given during 7-day Washout. Matching placebo administered once daily with food at 5 pm during the 28-day Second Treatment Intervention Period and the 7-day Second Taper Period. No treatment was given during Follow-up.
Period: First Treatment Intervention Period
Arm/Group | Placebo Followed by GEn 1200 mg/Day | GEn 1200 mg/Day Followed by Placebo
Started | 69 | 67
Completed | 64 | 66
Not Completed | 5 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: First Taper Period
Arm/Group | Placebo Followed by GEn 1200 mg/Day | GEn 1200 mg/Day Followed by Placebo
Started | 64 | 66
Completed | 61 | 65
Not Completed | 3 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Protocol Stopping Criteria Met | 0 | 1
Period: 1-Week Washout Period
Arm/Group | Placebo Followed by GEn 1200 mg/Day | GEn 1200 mg/Day Followed by Placebo
Started | 61 | 65
Completed | 59 | 64
Not Completed | 2 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0
Period: Second Treatment Intervention Period
Arm/Group | Placebo Followed by GEn 1200 mg/Day | GEn 1200 mg/Day Followed by Placebo
Started | 59 | 64
Completed | 53 | 61
Not Completed | 6 | 3
Not completed — Adverse Event | 4 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Second Taper Period
Arm/Group | Placebo Followed by GEn 1200 mg/Day | GEn 1200 mg/Day Followed by Placebo
Started | 53 | 61
Completed | 53 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants in the Intent-to-Treat (ITT) Population: All randomized participants who took at least one dose of study drug and had at least one post-baseline polysomnography (PSG) efficacy assessment
Arm/Group | All Participants in the Intent-to-Treat (ITT) Population
Number analyzed (Participants) | 131
Age Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristics were collected for all participants prior to the Baseline period and are summarized independent of treatment sequence. The ITT Population consisted of all randomized participants who took at least one dose of investigational product, and had at least one post-baseline polysomnography (PSG) sleep efficacy assessment.
  Years | 52.0 (12.70)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristics were collected for all participants prior to the Baseline period and are summarized independent of treatment sequence. The ITT Population consisted of all randomized participants who took at least one dose of investigational product, and had at least one post-baseline polysomnography (PSG) sleep efficacy assessment.
  Participants
    Female | 76
    Male | 55
Race/Ethnicity, Customized [Number; unit: participants] — Baseline characteristics were collected for all participants prior to the Baseline period and are summarized independent of treatment sequence. The ITT Population consisted of all randomized participants who took at least one dose of investigational product, and had at least one post-baseline polysomnography (PSG) sleep efficacy assessment.
  participants
    African American/African Heritage | 7
    American Indian or Alaska Native | 2
    Asian | 1
    White | 120
    Mixed Race | 1

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Wake Time During Sleep (WTDS) at Week 4/10 Measured by Polysomnography (PSG) (Sleep Study) Using Last Observation Carried Forward (LOCF)
Description: PSG is a comprehensive recording of the bio-physiological changes that occur during sleep. It is also known as a "sleep study" that monitors participants as they sleep or try to sleep. WTDS, defined as the total amount of time spent awake after falling asleep until the last awakening, was measured by PSG. Change from baseline was calculated as the Week 4 and Week 10 values minus the baseline value. Mean change from baseline was adjusted for treatment, pooled center, and period effects.
Time Frame: Baseline, Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: ITT Population: Of the 131 ITT participants, 2 and 6 participants did not take Placebo and GEn 1200 mg, respectively, in the second period. In addition, 6 placebo and 4 GEn 1200 participants did not have PSG data during the second intervention period and were therefore not included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: minutes
Groups:
- Placebo: Placebo once daily either in first intervention period or second intervention period
- GEn 1200 mg: GEn 1200 mg once daily either in first intervention period or second intervention period
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 123 | 121
minutes | -6.02 (4.986) | -32.02 (5.020)
Statistical Analysis 1: Comparison: Placebo vs GEn 1200 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Estimates were obtained using an ANCOVA model with period, group center, and treatment as fixed effects and participant as a random effect; Adjusted mean difference versus placebo = -26.00, 95% CI 2-sided [-35.64 to -16.36]

2. Secondary Outcome: Adjusted Mean Change From Baseline in Periodic Limb Movements Associated With Arousal (PLMAI) at Week 4/10 as Measured by Polysomnography Using LOCF
Description: PLMAI is defined as the number of Periodic Limb Movements (PLMs or involuntary jerks of the legs that cause a participant to arouse from sleep per hour of sleep). Change from baseline was calculated as the Week 4 and Week 10 values minus the baseline value. Mean change from baseline was adjusted for treatment, pooled center, and period effects.
Time Frame: Baseline, Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: limb movements per hour
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 123 | 121
limb movements per hour | -1.52 (0.892) | -4.59 (0.899)
Statistical Analysis 1: Comparison: Placebo vs GEn 1200 mg; Test type: Superiority or Other; p = 0.002, ANCOVA; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference versus placebo = -3.07, 95% CI 2-sided [-5.04 to -1.10]

3. Secondary Outcome: Adjusted Mean Change From Baseline in the International Restless Legs Rating Scale (IRLS) Total Score at Week 4/10 Using LOCF
Description: The IRLS is a measure of RLS disease severity. Ten items (individually scored from 0 to 4) are included that assess the impact of symptoms on participants' mood, daily life, and activities. The total scale score is a sum of all of the individual item scores and ranges from 0-40 points, with 40 being the most severe. The scale assesses symptoms over the week prior to measurement. Change from baseline was calculated as the Week 4 and Week 10 values minus the baseline value. Mean change from baseline was adjusted for treatment, pooled center, and period effects.
Time Frame: Baseline, Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: ITT Population: Of the 131 ITT participants, 2 and 6 participants did not take Placebo and GEn 1200 mg, respectively, in the second period. An additional 4 participants (2 in each treatment group) were excluded from the analysis due to missing/incomplete data.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 127 | 123
scores on a scale | -8.42 (0.713) | -14.99 (0.725)

4. Secondary Outcome: Adjusted Mean Change From Baseline in the Item 4 (Sleep Disturbance) Scores of the IRLS Rating Scale at Week 4/10 Using LOCF
Description: The IRLS is a measure of RLS disease severity. Item 4 of the IRLS evaluates RLS-related sleep impairment. It asks: "In the past week, how severe was your sleep disturbance due to your RLS symptoms?". The item is participant rated using a 5-point scale, where 0 is the absence of any sleep disturbance and 4 is very severe disturbance. Change from baseline was calculated as the Week 4 and Week 10 values minus the baseline value. Mean change from baseline was adjusted for treatment, pooled center, and period effects.
Time Frame: Baseline, Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 127 | 123
scores on a scale | -1.47 (0.092) | -2.27 (0.093)

5. Secondary Outcome: Adjusted Mean Change From Baseline in Time Spent in N1 Sleep as Measured by Polysomnography at Week 4/10 Using LOCF
Description: Stage N1 is considered "light sleep," during which participants drift in and out of sleep and can be awakened easily. In this stage, the eyes move slowly and muscle activity slows. This stage is sometimes referred to as "somnolence" or "drowsy sleep." Sudden twitches and hypnic jerks may be associated with the onset of sleep during N1. Change from baseline was calculated as the Week 4 and Week 10 values minus the baseline value. Mean change from baseline was adjusted for treatment, pooled center, and period effects.
Time Frame: Baseline, Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 123 | 121
minutes | -0.95 (1.508) | -6.19 (1.517)

6. Secondary Outcome: Adjusted Mean Change From Baseline in the Percentage of Total Sleep Time Spent in the N1 Sleep Stage at Week 4/10 Using LOCF
Description: Percentage of stage N1 sleep time was defined as the time spent in stage N1 sleep divided by total sleep time. Change from baseline was calculated as the Week 4 and Week 10 values minus the baseline value. Mean change from baseline was adjusted for treatment, pooled center, and period effects.
Time Frame: Baseline, Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of total sleep time
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 123 | 121
percentage of total sleep time | -0.23 (0.507) | -2.55 (0.511)

7. Secondary Outcome: Adjusted Mean Change From Baseline in Time Spent in the N2 Sleep Stage as Measured by Polysomnography at Week 4/10 Using LOCF
Description: In stage N2 of sleep, eye movement stops and brain waves become slower, with only an occasional burst of rapid brain waves. Participants may also experience spontaneous periods of muscle tone mixed with periods of muscle relaxation. During this stage, muscular activity, and conscious awareness of the external environment disappears. Change from baseline was calculated as the Week 4 and Week 10 values minus the baseline value. Mean change from baseline was adjusted for treatment, pooled center, and period effects.
Time Frame: Baseline, Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 123 | 121
minutes | 2.78 (4.528) | 22.95 (4.563)

8. Secondary Outcome: Adjusted Mean Change From Baseline in the Percentage of Total Sleep Time Spent in the N2 Sleep Stage at Week 4/10
Description: Percentage of stage N2 sleep time was defined as the time spent in stage N2 sleep divided by total sleep time. Change from baseline was calculated as the Week 4 and Week 10 values minus the baseline value. Mean change from baseline was adjusted for treatment, pooled center, and period effects.
Time Frame: Baseline, Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of total sleep time
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 123 | 121
percentage of total sleep time | 0.16 (0.808) | 0.64 (0.815)

9. Secondary Outcome: Mean Change From Baseline in the Total Time Spent in Stage N3 Sleep Time at Week 4/10 Measured by PSG Using LOCF
Description: Stage N3 is referred to as deep sleep; it is very difficult to wake a participant in this stage of sleep. In deep sleep, there is no eye movement or muscle activity. Change from baseline was calculated as the Week 4 and Week 10 values minus the baseline value. Mean change from baseline was adjusted for treatment, pooled center, and period effects.
Time Frame: Baseline, Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 123 | 121
minutes | 2.89 (2.351) | 15.02 (2.371)

10. Secondary Outcome: Adjusted Mean Change From Baseline in the Percentage of Total Sleep Time Spent in the N3 Sleep Stage at Week 4/10
Description: Percentage of stage N3 sleep time was defined as the time spent in stage N3 sleep divided by total sleep time. Change from baseline was calculated as the Week 4 and Week 10 values minus the baseline value. Mean change from baseline was adjusted for treatment, pooled center, and period effects.
Time Frame: Baseline, Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of total sleep time
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 123 | 121
percentage of total sleep time | 0.57 (0.559) | 2.62 (0.564)

11. Secondary Outcome: Adjusted Mean Change From Baseline in Time Spent in the REM (Rapid Eye Movement) Sleep Stage at Week 4/10 as Measured by Polysomnography Using LOCF
Description: In REM sleep, a participant's breathing becomes more rapid, irregular, and shallow; eyes jerk rapidly; and limb muscles are temporarily paralyzed. Brain waves during this stage increase to levels experienced when a person is awake. This is the stage when most dreams occur. Change from baseline was calculated as the Week 4 and Week 10 values minus the baseline value. Mean change from baseline was adjusted for treatment, pooled center, and period effects.
Time Frame: Baseline, Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 123 | 121
minutes | -1.21 (2.638) | 4.22 (2.659)

12. Secondary Outcome: Adjusted Mean Change From Baseline in the Percentage of Total Sleep Time Spent in the REM Sleep Stage at Week 4/10
Description: Percentage of stage REM sleep time was defined as the time spent in stage REM sleep divided by total sleep time. Change from baseline was calculated as the Week 4 and Week 10 values minus the baseline value. Mean change from baseline was adjusted for treatment, pooled center, and period effects.
Time Frame: Baseline, Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of total sleep time
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 123 | 121
percentage of total sleep time | -0.49 (0.582) | -0.71 (0.586)

13. Secondary Outcome: Adjusted Mean Change From Baseline in Periodic Limb Movements Causing Awakening (PLMAWI) at Week 4/10 as Measured by Polysomnography Using LOCF
Description: PLMAWI is defined as the number of PLMs (involuntary leg movements) that caused participants to wake up per hour of sleep. It is calculated by dividing the number of PLMs causing awakening by the total number of hours of sleep. Change from baseline was calculated as the Week 4 and Week 10 values minus the baseline value. Mean change from baseline was adjusted for treatment, pooled center, and period effects.
Time Frame: Baseline, Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: number of PLMs/total hours of sleep
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 123 | 121
number of PLMs/total hours of sleep | -0.08 (0.047) | -0.22 (0.048)

14. Secondary Outcome: Number of PLMAI Responders at Week 4/10 Using LOCF
Description: PLMAI is defined as the number of PLMs associated with arousal per hour of sleep. Participants with <=5 PLMAI were evaluated as responders.
Time Frame: Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 123 | 121
participants | 44 | 64

15. Secondary Outcome: Adjusted Mean Change From Baseline in Sleep Quality at Week 4/10 as Measured by the Subjective Post Sleep Diary (SPSD) Using LOCF
Description: Each day upon awakening, participants rated their overall sleep quality for the previous night on an 11-point scale (0=poor to 10=excellent) using the SPSD. Response to sleep quality was calculated for each visit by averaging the last 7 available diary days. Only participants with at least 4 days of diary data available (not in consecutive order) at any visit were included in the analysis. Change from baseline was calculated as the Week 4 and Week 10 values minus the baseline value. Mean change from baseline was adjusted for treatment, pooled center, and period effects.
Time Frame: Baseline, Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: ITT Population: The number of participants assessed varied due to missing/incomplete diary data.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 116 | 109
scores on a scale | 0.85 (0.141) | 1.95 (0.145)

16. Secondary Outcome: Adjusted Mean Change From Baseline in Participant's Ratings of Feeling Rested Upon Awakening as Measured by the Subjective Post Sleep Diary (SPSD) at Week 4/10 Using LOCF.
Description: Each day upon awakening, participants rated how rested they felt upon awakening on an 11-point scale (0=poor to 10=excellent) using the SPSD. Response to feeling rested upon awakening was calculated for each visit by averaging the last 7 available diary days. Only participants with at least 4 days of diary data available (not in consecutive order) at any visit were included in the analysis. Change from baseline was calculated as the Week 4 and Week 10 values minus the baseline value. Mean change from baseline was adjusted for treatment, pooled center, and period effects.
Time Frame: Baseline, Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: ITT Population: The number of participants assessed varied due to missing/incomplete diary data.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 116 | 109
scores on a scale | 0.83 (0.142) | 1.68 (0.146)

17. Secondary Outcome: Adjusted Mean Change From Baseline in the Number of Awakenings Measured Objectively by Polysomnography at Week 4/10 Using LOCF
Description: The number of awakenings was measured by PSG and is defined as the number of wake periods lasting at least 1 minute. Change from baseline was calculated as the Week 4 and Week 10 values minus the baseline value. Mean change from baseline was adjusted for treatment, pooled center, and period effects.
Time Frame: Baseline, Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: awakenings
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 123 | 121
awakenings | -0.56 (0.411) | -3.04 (0.414)

18. Secondary Outcome: Adjusted Mean Change From Baseline in the Self-reported Number of Hours Spent Awake During the Night (SPSD) Due to RLS at Week 4/10 Using LOCF
Description: Each day upon awakening, participants recorded, using the SPSD, the total number of hours spent awake the previous night due to RLS. Response to number of hours awake was calculated for each visit by averaging the last 7 available diary days. Only participants with at least 4 days of diary data available (not in consecutive order) at any visit were included in the analysis. Change from baseline was calculated as the Week 4 and Week 10 values minus the baseline value. Mean change from baseline was adjusted for treatment, pooled center, and period effects.
Time Frame: Baseline, Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: ITT Population: The number of participants assessed varied due to missing/incomplete diary data.
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 116 | 109
hours | -0.45 (0.064) | -0.56 (0.065)

19. Secondary Outcome: Number of Participants With no Self-reported Awakenings (SPSD) Due to RLS at Week 4/10 Using LOCF
Description: Each day upon awakening, participants recorded, using the SPSD, the number of awakenings due to RLS they experienced the previous night. Number of awakenings was calculated for each visit by averaging the last 7 available diary days. Only participants with at least 4 days of diary data available (not in consecutive order) at any visit were included in the analysis.
Time Frame: Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: ITT Population: The number of participants assessed varied due to missing/incomplete diary data.
Measure: Number; unit: participants
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 125 | 115
participants | 68 | 87

20. Secondary Outcome: Adjusted Mean Change From Baseline in the Total Sleep Time Measured by Polysomnography (PSG) at Week 4/10 Using LOCF
Description: Total sleep time is the number of minutes participants slept on average during the 8-hour polysomnography. Scoring of PSG data to yield measure of total sleep time was conducted at a central site in the United States. Change from baseline was calculated as the Week 4 and Week 10 values minus the baseline value. Mean change from baseline was adjusted for treatment, pooled center, and period effect.
Time Frame: Baseline, Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 123 | 121
minutes | 3.62 (5.572) | 36.32 (5.615)

21. Secondary Outcome: Adjusted Mean Change From Baseline in the Sleep Efficiency Measured by Polysomnography (PSG) at Week 4/10 Using LOCF
Description: Sleep efficiency is a percentage that is calculated by dividing total sleep time by the amount of time the participant was in bed during the PSG. Change from baseline was calculated as the Week 4 and Week 10 values minus the baseline value. Mean change from baseline was adjusted for treatment, pooled center, and period effect.
Time Frame: Baseline, Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: minutes/hour
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 123 | 121
minutes/hour | 0.76 (1.161) | 7.57 (1.170)

22. Secondary Outcome: Adjusted Mean Change From Baseline in the Wake After Sleep Onset (WASO) Measured by Polysomnography (PSG) at Week 4/10 Using LOCF.
Description: Wake After Sleep Onset (WASO) is defined as the total amount of time spent awake after falling asleep until the end of PSG recording. This endpoint is measured objectively by PSG. Change from baseline was calculated as the Week 4 and Week 10 values minus the baseline value. Mean change from baseline was adjusted for treatment, pooled center, and period effects
Time Frame: Baseline, Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 123 | 121
minutes | -3.76 (4.964) | -32.24 (5.002)

23. Secondary Outcome: Adjusted Mean Change From Baseline in the Suggested Immobilization Test (SIT) PLM Index at Week 4/10
Description: During the SIT, participants sat in bed with legs extended for 1 hour and were asked to rate their leg discomfort on a 100 millimeters visual analog scale every 5 minutes (score of 0-100, 0=none, higher numbers indicate more discomfort) and PLMs were assessed. The SIT-PLM Index is defined as the number of PLMs per hour during the SIT. Mean change from baseline was adjusted for treatment, pooled center, and period effects. Only results from SITs performed before a PSG assessment and of at least 60 minutes in length are included in the analysis.
Time Frame: Baseline, Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: ITT Population: The number of participants assessed varied due to missing/incomplete data.
Measure: Least Squares Mean (Standard Error); unit: number of PLMs per hour
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 119 | 117
number of PLMs per hour | -3.73 (7.394) | -30.52 (7.436)

24. Secondary Outcome: Adjusted Mean Change From Baseline in the SIT MDS (Mean Leg Discomfort Score), Mean of Scores From 0 to 60 Minutes, at Week 4/10
Description: During the SIT, participants sat in bed with legs extended for 1 hour and rated their leg discomfort on a visual analog scale every 5 minutes (range 0-100, 0=none, higher numbers indicate more discomfort). The SIT MDS is the average rating of leg discomfort during the specified time frame. Change from baseline was calculated as the Week 4 and Week 10 values minus the baseline value. Mean change from baseline was adjusted for treatment, pooled center, and period effects. Only results from SITs performed before a PSG assessment and of at least 60 minutes in length are included in the analysis.
Time Frame: Baseline, Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: ITT Population: The number of participants assessed varied due to missing/incomplete data.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 118 | 117
scores on a scale | -8.57 (2.136) | -21.24 (2.145)

25. Secondary Outcome: Number of Participants Who Responded Affirmatively to Each of the 4 Items of the Participant-completed Patient Global Impression of Therapy at Week 4/10 Using LOCF
Description: Each participant completed the participant-completed Patient Global Impression questionnaire at the end of each Treatment Period (Weeks 4 and 10) or Early Withdrawal. This instrument was developed to capture a participant's subjective assessment of therapy and is composed of the following 4 questions with dichotomous (Yes or No) responses: "Helped me sleep," "Helped me fall asleep faster," "Helped me sleep longer," and "Helped me get a better night's sleep."
Time Frame: Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: ITT Population: The number of participants assessed varied due to missing/incomplete data.
Measure: Number; unit: participants
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 123 | 118
participants
  Helped me sleep | 53 | 95
  Helped me fall asleep faster | 39 | 77
  Helped me sleep longer | 31 | 80
  Helped me get a better night's sleep | 50 | 89

26. Secondary Outcome: Adjusted Mean Change From Baseline in the Clinical Global Impression of Illness - Severity (CGI-S) Score at Week 4/10 Using LOCF
Description: The CGI-S scale allows the investigator to rate the severity of participants' illness considering their total clinical experience with the participant population being studied and based on all information available at the time of rating. The scale is rated from 1-7 (1=Normal, not at all ill; 7=Among the most extremely ill patients). Change from baseline was calculated as the Week 4 and Week 10 values minus the baseline value. Mean change from baseline was adjusted for treatment, pooled center, and period effects.
Time Frame: Baseline, Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: ITT Population: The number of participants assessed varied due to missing/incomplete data.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 121 | 118
scores on a scale | -1.18 (0.119) | -2.43 (0.121)

27. Secondary Outcome: Number of Participants Who Were Defined as Clinical Global Impression of Illness (CGI-I) Scale "Responders" at Week 4/10 Using LOCF
Description: The CGI-I scale allows the investigator to rate the participant's global improvement or worsening compared with the condition at baseline (i.e., Day 1), and whether or not the change is thought to be due to treatment with study medication. The scale is rated from 1-7 (1=Very much improved to 7=Very much worse). Participants with a score of 1 ("Very much improved") or 2 ("Much improved") are considered to be responders.
Time Frame: Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: ITT Population: The number of participants assessed varied due to missing/incomplete data.
Measure: Number; unit: participants
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 127 | 123
participants | 46 | 91

28. Secondary Outcome: Number of Participants Who Self-reported "Very Satisfied" or "Satisfied" With the Investigational Product at Week 4/10 Using LOCF
Description: Participant satisfaction with RLS medication was captured on a seven-point ordinal scale. The scale asked "Overall, how satisfied are you with the medication you received for the treatment of your RLS symptoms during the study." The participant responses ranged from 1 ("Very satisfied") to 7 ("Very dissatisfied"). A "satisfied" response was scored a 2.
Time Frame: Week 4/10 (representing the last week of each intervention period, i.e. Weeks 4 and 10)
Population: ITT Population: The number of participants assessed varied due to missing/incomplete data.
Measure: Number; unit: participants
Arm/Group | Placebo | GEn 1200 mg
Number analyzed (Participants) | 122 | 118
participants
  Very Satisfied | 22 | 38
  Satisfied | 23 | 35

ADVERSE EVENTS:
Time Frame: Adverse event (AE) and serious adverse event (SAE) collection started immediately following informed consent and continued throughout the study (up to Week 12).
Description: AEs and SAEs were presented for the Safety Population, defined as all participants who were randomized and took at least one dose of investigational product. Participants were assigned to a treatment group within the Safety Population if they took at least one dose of that treatment (i.e., in that treatment period).
Groups:
- Placebo: Participants who took at least one dose of placebo in either the first intervention period or the second intervention period. Of the 136 participants in the Safety Population, 132 took at least one dose of placebo.
- GEn 1200 mg: Participants who took at least one dose of GEn 1200 mg in either the first intervention period or the second intervention period. Of the 136 participants in the Safety Population, 127 took at least one dose of GEn 1200 mg.
Arm/Group | Placebo | GEn 1200 mg
Serious Adverse Events (participants affected / at risk) | 0/132 | 2/127
Other Adverse Events (participants affected / at risk) | 27/132 | 54/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=132) | GEn 1200 mg (N=127)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=132) | GEn 1200 mg (N=127)
Dizziness (Nervous system disorders) | 3 (3) | 26 (26)
Headache (Nervous system disorders) | 9 (9) | 11 (11)
Somnolence (Nervous system disorders) | 2 (2) | 16 (16)
Dry mouth (Gastrointestinal disorders) | 5 (5) | 6 (6)
Nausea (Gastrointestinal disorders) | 5 (5) | 6 (6)
Constipation (Gastrointestinal disorders) | 4 (4) | 6 (6)
Nasopharyngitis (Immune system disorders) | 4 (4) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.